CLINICAL TRIAL: NCT04069520
Title: Neuroplastic Mechanisms Underlying Augmented Neuromuscular Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Greg Myer, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00001772; 1R01AR076153 (NIH); 2019-0245 (Other: CCHMC Institutional Review Board)
Record Dates: First submitted 2019-07-09; First posted 2019-08-28 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aNMT Biofeedback (Experimental): Participants randomized to receive a neuromuscular training intervention that incorporates biofeedback training.
  Interventions: Other: aNMT Biofeedback
- Sham Biofeedback (Sham Comparator): Participants randomized to receive a neuromuscular training intervention with sham feedback training.
  Interventions: Other: Sham Biofeedback

INTERVENTIONS:
Other: aNMT Biofeedback — aNMT biofeedback is created by calculating kinematic and kinetic data in real-time from the athlete's own movements. These values determine real-time transformations of the stimulus shape the athlete views via augmented-reality (AR) glasses during movement performance. The athlete's task is to move so as to create ("animate") a particular stimulus shape that corresponds to desired values of the biomechanical parameters targeted by the intervention. The aNMT biofeedback occurs during neuromuscular training sessions. The neuromuscular training is a 18 session, pre-season training program occurring over 6 weeks.
  Arms: aNMT Biofeedback
Other: Sham Biofeedback — Sham biofeedback provides a similar phenomenological experience to aNMT biofeedback for athletes-both groups experience a shape that changes with their movements-but the sham biofeedback will not provide usable information to modify movement parameters during critical movement phases. The sham biofeedback occurs during neuromuscular training sessions. The neuromuscular training is a 18 session, pre-season training program occurring over 6 weeks.
  Arms: Sham Biofeedback

SUMMARY:
The purpose of this study is to determine the neural mechanisms of augmented neuromuscular training (aNMT). Participants will complete a 6-week course of neuromuscular training with either aNMT biofeedback or sham biofeedback. An MRI will be performed before and after the training program.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury is a common and debilitating knee injury affecting over 350,000 children or young adults each year, drastically reducing their chances for an active and healthy life. Annual direct costs exceed $13 billion, and the long-term indirect costs far exceed that figure, as ACL injury is also linked to accelerated development of disabling osteoarthritis within a few years after injury. The National Public Health Agenda for Osteoarthritis recommends expanding and refining evidence-based ACL injury prevention to reduce this burden. The investigators have identified modifiable risk factors that predict ACL injury in young female athletes. This neuromuscular training targets those factors and shows statistical efficacy in high-risk athletes, but meaningful transfer of low-risk mechanics to the field of play has been limited, as current approaches are not yet decreasing national ACL injury rates in young female athletes. The key gap is how to target mechanisms that allow transfer of risk-reducing motor control strategies from the intervention to the athletic field. The mechanisms that ultimately make such transfer possible are neural, but thus far injury prevention training focusing on neuromuscular control has not utilized neural outcomes. The investigators published and new preliminary data on neuroplasticity related to injury and neuromuscular training demonstrate the proficiency to capture these neural outcomes and future capability to target these neural mechanisms to improve the rate of motor transfer. The data support this proposal's central hypothesis that increased sensory, visual and motor planning activity to improve motor cortex efficiency is the neural mechanism of adaptation transfer to realistic scenarios. The ability to target the neural mechanisms to increase risk-reducing motor transfer from the clinic to the world could revolutionize ACL injury prevention. The transformative, positive impact of such innovative strategies will enhance the delivery of biofeedback to optimize training and increase the potential for sport transfer. This contribution will be significant for ACL injury prevention and associated long-term sequelae in young females. This unique opportunity to enhance ACL injury prevention by targeting neural mechanisms of neuromuscular adaptation and transfer will reduce the incidence of injuries that cause costly and long-term disabling osteoarthritis.

Participants from the parent study "Real-time Sensorimotor Feedback for Injury Prevention Assessed in Virtual Reality" will be eligible to participate in this study. In the parent study, participants are randomized to receive augmented neuromuscular training (aNMT) or sham biofeedback training that will be evaluated using 3D biomechanical assessments. Enrolled participants into the current ancillary project will complete MRI testing before and after the study training program. The MRI protocol will include high resolution T1-weighted 3D images, motor task-based functional magnetic resonance imaging (fMRI). The fMRI tasks will be focused on motor function, participants will be asked to complete lower extremity movements including knee flexion and extension and a combined hip and knee flexion and extension.

ELIGIBILITY:
Inclusion Criteria:

- enrolled in parent study "Real-time Sensorimotor Feedback for Injury Prevention Assessed in Virtual Reality"

Exclusion Criteria:

- contraindications to MRI scan

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Healthcare Sports Performance And Research Center (SPARC), Flowery Branch, Georgia
  - Cincinnati Childrens Hospital Medical Center (CCHMC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- aNMT Biofeedback: Participants randomized to receive a neuromuscular training intervention that incorporates aNMT biofeedback training.
  aNMT Biofeedback: aNMT biofeedback is created by calculating kinematic and kinetic data in real-time from the athlete's own movements. These values determine real-time transformations of the stimulus shape the athlete views via augmented-reality (AR) glasses during movement performance. The athlete's task is to move so as to create ("animate") a particular stimulus shape that corresponds to desired values of the biomechanical parameters targeted by the intervention. The aNMT biofeedback occurs during neuromuscular training sessions. The neuromuscular training is a 18 session, pre-season training program occurring over 6 weeks.
Period: Overall Study
Arm/Group | aNMT Biofeedback | Sham Biofeedback
Started | 48 | 45
Completed | 46 | 40
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Prior Injury | 1 | 0
Not completed — Orthodontia | 1 | 0
Not completed — Cut from team | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- aNMT Biofeedback: Female basketball, soccer and volleyball player enrolled in high school or club teams were randomized to receive a neuromuscular training intervention that incorporates biofeedback training.
- Sham Biofeedback: Female basketball, soccer and volleyball players enrolled in high school or club teams were randomized to receive a neuromuscular training intervention that incorporates Sham biofeedback training.
- Total: Total of all reporting groups
Arm/Group | aNMT Biofeedback | Sham Biofeedback | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.39 (1.22) | 15.55 (1.30) | 15.47 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 45 | 93
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 39 | 35 | 74
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 4 | 6 | 10
  White | 31 | 26 | 57
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 48 | 45 | 93

OUTCOME MEASURES:

1. Primary Outcome: Neural Mechanisms for Injury-resistant Movement Pattern Acquisition
Description: Sensorimotor brain activity was measured in task-based fMRI (% Blood Oxygen Level Dependent (BOLD) Signal change of knee sensorimotor network regions from baseline between rest and move blocks at each respective time point- the standard measure to determine brain activity during a condition is to contrast to rest to remove confounds make the data interpretable across conditions and individuals) and was associated with knee joint biomechanics (knee sagittal and frontal plane angle and moments) captured during landing task during standard laboratory landing assessment pre- and post-intervention.
Time Frame: Baseline (pre-training testing), Week 7 (post-training testing)
Population: Number of participants at week 7 post-training includes subjects that were able to attend and complete the visit.
Measure: Mean (Standard Deviation); unit: % BOLD Signal change
Arm/Group | aNMT Biofeedback | Sham Biofeedback
Number analyzed (Participants) | 48 | 45
% BOLD Signal change
  Baseline (pre-training testing) | 0.28 (0.11) | 0.26 (0.17)
  Week 7 (post-training testing): number analyzed (Participants) | 46 | 40
  Week 7 (post-training testing) | 0.26 (0.17) | 0.21 (0.10)

2. Primary Outcome: Knee Joint Biomechanics During Landing Task
Description: Knee joint biomechanics (knee angle) captured during a standard laboratory landing task assessment was reported pre- and post-intervention. The degree of knee angle is the peak knee flexion angle during drop vertical jump landing.
Time Frame: Baseline (pre-training testing), Week 7 (post-training testing)
Population: Number of participants at week 7 post-training includes subjects that were able to attend and complete the visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | aNMT Biofeedback | Sham Biofeedback
Number analyzed (Participants) | 48 | 45
Degrees
  Knee angle at Baseline (pre-training testing) | 83.49 (10.00) | 80.50 (9.77)
  Knee angle at Week 7 (post-training testing): number analyzed (Participants) | 46 | 40
  Knee angle at Week 7 (post-training testing) | 86.06 (10.81) | 83.48 (10.36)

3. Secondary Outcome: Neural Mechanisms for Injury-resistant Movement Pattern Transfer to VR-simulated Sport
Description: Sensorimotor brain activity during task-based fMRI (% Blood Oxygen Level Dependent (BOLD) Signal change of knee sensorimotor network regions from baseline between rest and move blocks at each respective time point- the standard measure to determine brain activity during a condition is to contrast to rest to remove confounds make the data interpretable across conditions and individuals) was assessed and compared to biomechanical movement patterns (knee angle) measured during VR-simulated sport.
Time Frame: Baseline (pre-training testing), Week 7 (post-training testing)
Population: Number of participants at week 7 post-training includes subjects that were able to attend and complete the visit.
Measure: Mean (Standard Deviation); unit: % of BOLD signal change
Arm/Group | aNMT Biofeedback | Sham Biofeedback
Number analyzed (Participants) | 48 | 45
% of BOLD signal change
  Baseline (pre-training testing) | 0.31 (0.14) | 0.26 (0.13)
  Week 7 (post-training testing): number analyzed (Participants) | 46 | 40
  Week 7 (post-training testing) | 0.26 (0.13) | 0.31 (0.11)

4. Secondary Outcome: Knee Joint Biomechanics During VR-simulated Sport
Description: Biomechanical movement patterns (knee angle) were measured during VR-simulated sport at pre- and post-intervention. The degree of knee angle is the peak knee flexion angle during a sport specific landing task.
Time Frame: Baseline (pre-training testing), Week 7 (post-training testing)
Population: Number of participants at week 7 post-training includes subjects that were able to attend and complete the visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | aNMT Biofeedback | Sham Biofeedback
Number analyzed (Participants) | 48 | 45
Degrees
  Knee angle at Baseline (pre-training testing) | 68.43 (10.93) | 68.93 (12.10)
  Knee angle at Week 7 (post-training testing): number analyzed (Participants) | 46 | 40
  Knee angle at Week 7 (post-training testing) | 73.27 (12.76) | 71.89 (12.09)

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post-intervention
Arm/Group | aNMT Biofeedback | Sham Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 0/48 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04069520/Prot_003.pdf
  • Informed Consent Form (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04069520/ICF_004.pdf